CLINICAL TRIAL: NCT03566758
Title: The Association Between Muscle Mass and Nutritional Risk by COAST in Older Adults
Brief Title: Muscle Mass and Nutritional Risk in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201801247
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the COAST (comprehensive older adult screening tool) to muscle mass as determined by BIA (bioelectric impedance analysis) and thus, determine if the COAST is a valid predictor of muscle loss in older adults. This study follows a comparison of COAST to MNA and will further test the validity of the COAST nutrition screening tool.

DETAILED DESCRIPTION:
The association between muscle mass, as determined by BIA (bioelectric impedance analysis), and the recently developed COAST (Comprehensive Older Adult Screening Tool) has not been studied. Therefore, the main objective of this study is to test the correlations between muscle mass, measured by BIA, and COAST. The population to be studied will be older adults (n=150). Participants will be included if they are 60 years or older, willing to have weight, height, handgrip and body composition measured, willing to provided demographic information and answer questions related to their nutritional and health status. Individuals will be excluded if they have had recent surgery to the hands, severe rheumatoid arthritis in both hands or have a pacemaker or other implanted device. Participants will be recruited from community groups in Florida. Participants muscle mass will be measured using BIA. Also, their handgrip strength will be tested using a dynamometer. Weight and height will be measured and demographic information will be collected. In addition, the participants will be given COAST (5 questions related to their nutritional and health status). The associations among BIA, handgrip strength and the COAST will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 60 -100 years of age
* willing to weight, height, handgrip and body composition measured, willing to provide demographic information and answer questions related to their nutritional and health status

Exclusion Criteria:

* recent surgery to the hands, severe rheumatoid arthritis in both hands or have a pacemaker or other implanted device.

Ages: 60 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Older adults
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
COAST (Comprehensive Older Adult Screening Tool) score | baseline only
  Ability of the COAST score to predict depleted muscle mass. A five question survey, scored from 0 to 8 points; 8 being the maximum score.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No